CLINICAL TRIAL: NCT01064999
Title: An Open Label, Randomized, Multi-center, Phase II/III Trial of High Intensity Versus Low Intensity Neoadjuvant Chemoradiotherapy With Intensity-modified Radiation Therapy (IMRT) in Local Advanced Rectal Cancer
Brief Title: A Trial of High Intensity Versus Low Intensity Neoadjuvant Chemoradiotherapy in Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Collaborators: Zhejiang Cancer Hospital (Other); First People Hospital of Zhejiang (Unknown); RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Division Head, Division of Radiation Oncology,Cancer Hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-002
Record Dates: First submitted 2010-02-05; First posted 2010-02-09 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Rectal Cancer
Keywords: Neoadjuvant chemotherapy; locally advanced rectal cancer; intensity-modulated radiation therapy; pathological complete response
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High intensity group (Experimental): (RT 55Gy + CapOx) + a cycle of Xelox + Surgery
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Radiation: Radiotherapy; Procedure: Surgery
- Low instensity group (Active Comparator): (RT 50Gy + CapOx) + Surgery
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Radiation: Radiotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: Oxaliplatin — CRT:50mg/m2,IV,weekly*5 cycle CT: 130mg/m2,IV,d1,q 21 day
Drug: Capecitabine — CRT:625mg/m2,bid,d1-5,q week RT:1000mg/m2,bid,d1-14,q 3 weeks
Radiation: Radiotherapy — High intensity group:55Gy Low intensity group:50Gy
Procedure: Surgery — Lower anterior resection or abdominoperineal resection

SUMMARY:
Neoadjuvant chemoradiotherapy (CRT) has been the standard therapy for local advanced rectal cancer. Pathological complete response (pCR) is an important prognostic factor for local control and survival. A high intensity CRT increases not only the pCR rate, but also toxicity, especially diarrhea. Compared with traditional RT technique, intensity-modified radiation therapy (IMRT) can decrease the toxicity of diarrhea because of low volume of high dose for small bowel. Therefore, IMRT technique provides an opportunity to improve the dose intensity of neoadjuvant CRT. The investigators hypothesize that a higher treatment dose induces a high rate of pCR and design a two-arm trial. in this trial, low intensity CRT includes the whole pelvic irradiation of 50Gy together with Oxaliplatin and Capecitabine weekly. While in high intensity group, additional concomitant 5Gy for primary tumor and a cycle of Xelox are prescribed. All patients will receive a total mesorectal excision (TME) 8 weeks after CRT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal adenocarcinoma
* Clinical staged T3/4 or any node-positive disease
* Age: 18-75 years
* Karnofsky Performance Status > 80
* Adequate bone marrow reserve, renal and hepatic functions
* Without previous antitumoural chemotherapy
* No evidence of metastatic disease
* Written informed consent before randomization

Exclusion Criteria:

* Previous pelvis radiotherapy.
* Previous antitumoural chemotherapy
* Clinically significant internal disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-03 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
the rate of pathological complete response (pCR) | within 14days after surgery
toxicity | every week during radiotherapy

SECONDARY OUTCOMES:
local recurrence | every half year after surgery
disease-free survival | every half year after surgery
overall survival | every half year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang J, Guan Y, Gu W, Yan S, Zhou J, Huang D, Tong T, Li C, Cai S, Zhang Z, Zhu J. Long-course neoadjuvant chemoradiotherapy with versus without a concomitant boost in locally advanced rectal cancer: a randomized, multicenter, phase II trial (FDRT-002). Radiat Oncol. 2019 Nov 29;14(1):215. doi: 10.1186/s13014-019-1420-z. PMID 31783766